CLINICAL TRIAL: NCT03046758
Title: The Safety and Pharmacokinetics of Intraperitoneal Administration of Granulocyte-macrophage Colony-stimulating Factor, Fosfomycin, and Metronidazole in Patients Undergoing Appendectomy for Uncomplicated Appendicitis
Brief Title: The Safety and Pharmacokinetics of Intraperitoneal Administration in Patients Undergoing Appendectomy for Uncomplicated Appendicitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Collaborators: Jacob Rosenberg (Sponsor) (Unknown); Barbara Juliane Holzknecht (Investigator) (Unknown); Magnus Arpi (Investigator) (Unknown); Johan Juhl Weisser (Partner, data analysis) (Unknown)
Responsible Party: Principal Investigator, Siv Fonnes, Principal Investigator, Herlev Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEH-SF-01
Record Dates: First submitted 2017-02-02; First posted 2017-02-08 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Metronidazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants (Experimental)
  Interventions: Drug: A combination of fosfomycin, metronidazole and GM-CSF i.p.

INTERVENTIONS:
Drug: A combination of fosfomycin, metronidazole and GM-CSF i.p. — All drugs will be administered together intraperitoneally at the end of the surgery after the appendix has been removed.

SUMMARY:
The objective of this trial is to evaluate the safety of the intraperitoneal administration of the combination of fosfomycin, metronidazole, and granulocyte-macrophage colony-stimulating factor (GM-CSF) in patients undergoing surgery for uncomplicated appendicitis. Further, in a sub-trial the aim is to investigate the plasma concentrations of fosfomycin and metronidazole after intraperitoneal administration.

ELIGIBILITY:
Inclusion Criteria:

* Men ≥18 years old
* Suspicion of acute appendicitis and planned for diagnostic laparoscopy and eventual appendectomy
* Written informed consent after written and verbal information

Exclusion Criteria:

* Cannot understand, read or speak Danish
* Previous allergic reaction to fosfomycin, metronidazole, or GM-CSF
* Perforated appendicitis (diagnosed either during surgery or at a preoperative computer tomography (CT) scan)
* Diagnostic laparoscopy revealing normal appendix not requiring an appendectomy
* Other intra-abdominal pathology requiring surgical intervention (diagnosed either during surgery or at a preoperative CT-scan)
* Known renal or hepatic disease or biochemical evidence at the time of admission
* Known autoimmune disease or other chronic inflammation
* Known hematologic disease or cancer
* Previous abdominal surgery (either laparoscopic or open surgery)
* Daily use or use of medication one week prior to or during the trial period apart from painkillers such as paracetamol, ibuprofen, tramadol, and morphine as well as drugs needed for anaesthesia, thrombosis prophylaxis, and nausea. Limitations for antibiotics are defined below
* Use of other antimicrobial agents than the trial treatment one month before until 24 hours after the trial treatment
* Participant in another drug trial one month prior to the date of the surgery
* Body mass index ≥35 kg/m2
* Weekly intake of alcohol >14 units, where one unit corresponds to 12 g alcohol

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2017-12-07 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
Main trial (14 patients): Drop of white blood cell counts | 4 hours (± 30 minutes)
  The safety of intraperitoneal administration is evaluated through the white blood cell counts 4 hours (± 30 minutes) postoperatively. A toxic effect is defined by a drop below the lower reference range.
Sub-trial (8 patients): The pharmacokinetics of fosfomycin. | Until 24 hours after surgery ±4 hours.
  The plasma concentrations of fosfomycin over time are measured with high-performance liquid chromatography mass spectrometry (HPLC-MS) until 24 hours after surgery ±4 hours.

SECONDARY OUTCOMES:
Main trial (14 patients): Biochemical markers | 4 hours ±30 minutes postoperatively.
  A standard panel of blood samples (e.g. white blood cell differential count, inflammation marker C-reactive protein (CRP), kidney function tests, liver function tests, and electrolytes) are analysed at admission (baseline) and 4 hours ±30 minutes postoperatively, these markers are compared.
Main trial (14 patients): Blood pressure | Until 12 hours ±30 minutes.
  Blood pressure in mmHg is measured perioperatively (baseline, 5 minutes, 10 minutes and 15 minutes after the trial treatment has been administered) and postoperatively (4 and 12 hours ±30 minutes after the trial treatment has been administered).
Main trial (14 patients): Pulse | Until 12 hours ±30 minutes.
  Pulse in beats per minute is measured perioperatively (baseline, 5 minutes, 10 minutes and 15 minutes after the trial treatment has been administered) and postoperatively (4 and 12 hours ±30 minutes after the trial treatment has been administered).
Main trial (14 patients): Frequency of respiration | Until 12 hours ±30 minutes.
  Frequency of respiration in breaths per minute is measured perioperatively (baseline, 5 minutes, 10 minutes and 15 minutes after the trial treatment has been administered) and postoperatively (4 and 12 hours ±30 minutes after the trial treatment has been administered).
Main trial (14 patients): Peripheral saturation | Until 12 hours ±30 minutes.
  Peripheral saturation of oxygen in percent is measured perioperatively (baseline, 5 minutes, 10 minutes and 15 minutes after the trial treatment has been administered) and postoperatively (4 and 12 hours ±30 minutes after the trial treatment has been administered).
Main trial (14 patients): Temperature | Until 12 hours ±30 minutes.
  Temperature in degrees Celsius is measured perioperatively (baseline, 5 minutes, 10 minutes and 15 minutes after the trial treatment has been administered) and postoperatively (4 and 12 hours ±30 minutes after the trial treatment has been administered).
Main trial (14 patients): Length of stay. | Until 30 days postoperatively.
  Length of stay in hours postoperatively (minimum length of stay: 12 hours but information on length of stay is collected until 30 days postoperatively).
Main trial (14 patients): Length of stay. | Until 30 days postoperatively.
  Length of stay in hours postoperatively (minimum 12 hours).
Main trial (14 patients): Side effects | 10 days postoperatively ±1 day.
  Side effects are evaluated through an objective examination and questions about changes 12 hours ±30 minutes and 10 days postoperatively ±1 day.
Main trial (14 patients): Adverse events | Until 30 days postoperatively.
  Adverse events are registered from the surgery until 30 days postoperatively through medical records and contact with the participant by telephone.
Sub-trial (8 patients): The pharmacokinetics of metronidazole. | Until 24 hours after surgery ±4 hours.
  The plasma concentrations of metronidazole over time are measured with HPLC-MS until 24 hours after surgery ±4 hours.
Sub-trial (8 patients): Microbiological flora and susceptibility | Until 30 days postoperatively.
  The microbiological flora and susceptibility of specimens collected during the surgery from the abdominal excess fluid and/or swab from the appendices are investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Siv Fonnes, MD, Principal Investigator — Center for Perioperative Optimization, Department of Surgery, Herlev Hospital
Locations (1):
- Department of Surgery, Herlev Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Fonnes S, Holzknecht BJ, Arpi M, Rosenberg J. Intraperitoneal administration of fosfomycin, metronidazole, and granulocyte-macrophage colony-stimulating factor in patients undergoing appendectomy is safe: a phase II clinical trial. Sci Rep. 2019 Apr 30;9(1):6727. doi: 10.1038/s41598-019-43151-4. PMID 31040341
- See also: Link to the article regarding the safety (open access) — https://www.nature.com/articles/s41598-019-43151-4